CLINICAL TRIAL: NCT05806333
Title: Diagnostic Performance of [18F]FAPI PET/CT in Suspicious Focal Liver Lesions Without FDG Avidity
Brief Title: [18F]FAPI PET/CT in Suspicious Focal Liver Lesions Without FDG Avidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Ji Bin, PHD, Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ChinaJapanUH
Record Dates: First submitted 2023-03-08; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- suspicious focal liver mass without FDG avidity (Experimental): Experimental: 18F-FAPI PET/CT Imaging was performed 30-60 minutes after injection of 2-4mci 68Ga-FAPI tracer
  Interventions: Diagnostic Test: FAPI PET

INTERVENTIONS:
Diagnostic Test: FAPI PET — Drug: 18F-FAPI 18F-FAPI were injected into the patients before the PET/CT scans

SUMMARY:
Fibroblast activation protein (FAP) is a serine protease that belongs to the dipeptidyl peptidase-IV (DPP-IV) family located in fbroblast membranes. FAP is overexpressed in the cancer-associated fbroblasts (CAFs) of 90% of epithelial carcinomas, including primary and metastatic liver cancer. We aim to conduct a prospective study to investigate the diagnostic perfoemance of 18F-FAPI PET/CT in evaluating suspicious liver mass without FDG avidity.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is a serine protease that belongs to the dipeptidyl peptidase-IV (DPP-IV) family located in fbroblast membranes. FAP is overexpressed in the cancer-associated fbroblasts (CAFs) of 90% of epithelial carcinomas, including primary and metastatic liver cancer. Therefore, FAP-targeted radiopharmaceuticals can be considered a promising approach for visualizing CAFs. CAFs are crucial components of the tumor stroma, promote the growth of cancer cells, and are associated with poor prognosis. Currently, 18F-labelled fbroblast activation protein inhibitor 18F-FAPI has shown promising diagnostic value in many types of tumors, especially those in which are not avid for 18F-FDF , and several studies have demonstrated that 18F-FAPI PET/CT is superior to 18F-FDG PET/CT for detecting liver cancer and has lower tracer uptake in normal liver tissue. We aim to conduct a prospective study to investigate the diagnostic performance of 18F-FAPI PET/CT in evaluating suspicious liver mass without FDG avidity.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected liver malignant lesions based on traditional diagnostic imaging (CT or MRI or ultrasound) and clinical symptoms;
* patients underwent [18F]FDG PET/CT with negative findings (suspicious primary and/or metastatic lesions were hypo- or isometabolic on [18F]FDG PET/CT);
* patients who agreed to undergo [18F]FAPI PET/CT scans within 1 week.

Exclusion Criteria:

* pregnancy;
* age<18 years old;
* patients with chemo/radio/targeted therapy before scanning;
* inability to provide informed consent (signed by participant, parent, or legal representative).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of FAPI PET | 1 year
  Sensitivity and specificity in detecting liver cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bin Ji, Principal Investigator — China-Japan Union Hospital, Jilin University
Locations (1):
- China-Japan Union Hospital, Changchun, Jilin, China